CLINICAL TRIAL: NCT01513525
Title: A Randomised, Open-label, Single Centre, Three Period Cross-over Trial in Healthy Subjects Comparing the Pharmacokinetic Profiles After Single Dose Administration of Liraglutide at Three Different Injection Sites
Brief Title: Comparison of Liraglutide Injected at Three Different Injection Sites in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN2211-1745; 2006-004670-27 (EudraCT Number)
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Abdomen (Experimental)
  Interventions: Drug: liraglutide
- Thigh (Experimental)
  Interventions: Drug: liraglutide
- Upper arm (Experimental)
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Single dose of 0.60 mg administered subcutaneously in three different injection sites on three separate dosing visits

SUMMARY:
This trial is conducted in Europe. the aim of this trial is to compare the pharmacokinetic profile of liraglutide between administrations in the thigh versus the abdomen and between administrations in the upper arm versus the abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Good general health as judged by the Investigator based on medical history, physical examination including 12-lead ECG (electrocardiogram), vital signs and blood and urinary laboratory assessments
* BMI (Body Mass Index): 18.5-27.5 kg/m^2, both inclusive

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods as required by local law or practice
* The receipt of any investigational drug within 3 months prior to this trial
* History of any clinically significant renal, hepatic, cardiovascular, pulmonary, gastrointestinal, metabolic, endocrine, haematological, neurological, psychiatric disease or other major disorders that may interfere with the objectives of the trial, as judged by the Investigator
* Impaired renal function
* Active hepatitis B and/or active hepatitis C
* Positive human immunodeficiency virus (HIV) antibodies
* Use of any prescription or non-prescription medication, except for paracetamol and vitamins
* History of alcoholism or drug abuse during the last 12 months.
* Smoking
* Habitual excessive consumption of methylxanthine-containing (theophylline, caffeine or theobromine) beverages and foods (coffee, tea, soft drinks such as red bull, cola, chocolate) as judged by the Investigator
* Excessive consumption of a diet deviating from a normal diet as judged by the Investigator
* Blood donation within the last 3 months
* Plasma donation within the last month

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2007-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Area under the Curve (AUC) of liraglutide for each injection site

SECONDARY OUTCOMES:
AUC
Cmax, maximum concentration
tmax, time to maximum concentration
t½, terminal half-life
Terminal elimination rate constant
Relative Bioavailability
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Kapitza C, Zdravkovic M, Zijlstra E, Segel S, Heise T, Flint A. Effect of three different injection sites on the pharmacokinetics of the once-daily human GLP-1 analogue liraglutide. J Clin Pharmacol. 2011 Jun;51(6):951-5. doi: 10.1177/0091270010374474. Epub 2010 Jul 29. No abstract available. PMID 20671294
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com